CLINICAL TRIAL: NCT04405427
Title: A Comparison of the Therapeutic Effect Between Head-point Acupuncture and Conventional Body Acupuncture on Insomnia: A Randomized Controlled Case Study
Brief Title: A Comparison of the Therapeutic Effect Between Head-point Acupuncture and Conventional Body Acupuncture on Insomnia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 201900496A3
Record Dates: First submitted 2020-05-24; First posted 2020-05-28 (Actual); Last update posted 2020-08-25 (Actual); Status verified 2020-05

CONDITIONS: Sleep Initiation and Maintenance Disorders
Keywords: acupuncture; primary insomnia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- head acupoints acupuncture (Experimental): Acupuncture treatment for 12 acupoints on both sides of the head
  Interventions: Procedure: head acupoints acupuncture
- body acupoints acupuncture (Active Comparator): Acupuncture treatment for 12 acupoints on both sides of the body
  Interventions: Procedure: body acupoints acupuncture

INTERVENTIONS:
Procedure: head acupoints acupuncture — The participants will undergo GV20, EX-HN-1, GV21, GV22, GV23, GV24, GV29, and GB13 head acupoints aupunture treatment 3 times/ 1 week for 4 weeks.
  Arms: head acupoints acupuncture
Procedure: body acupoints acupuncture — The participants will undergo HT7, PC6, SP6, ST36, KI3, and LR3 body acupoints acupunture treatment 3 time/1 week for 4 weeks.
  Arms: body acupoints acupuncture

SUMMARY:
The investigators will conduct a single-center, and randomized controlled cases study. A total of 120 participants with insomnia will be enrolled. The aim of the study is to compare the therapeutic effect between head-acupoints acupuncture and body-acupoints acupuncture on Insomnia.

DETAILED DESCRIPTION:
The investigators will conduct a single-center, and randomized controlled cases study. A total of 120 participants with insomnia will be enrolled, and randomly assigned into two groups, 60 of them are the head-acupoints acupuncture group, who will receive GV20, EX-HN-1, GV21, GV22, GV23, GV24, GV29, and bilateral GB13 head-acupoints acupuncture treatment, and 60 of them are the body-acupoints acupuncture group, who will receive bilateral HT7, PC6, SP6, ST36, KI3, LR3 body-acupoints acupuncture treatment for 4 weeks.

The primary outcomes of therapeutic effect on insomnia are changes of the Pittsburgh Sleep Quality Index (PSQI), Epworth Sleepiness Scale (ESS), and the Hospital Anxiety and Depression Scale (HADS).The time frame of the three primary outcomes are: baseline week 0, week 2, week 4 and week 6.

The secondary outcomes of therapeutic effect on insomnia are sleep parameters including sleep efficiency (SE), sleep awakenings (SA) and total sleep time (TST) recorded by the actigraphy (time frame: baseline week 0, week 2, week 4 and week 6), as well as the heart rate viability(HRV) recorded by the ECG monitor (time frame: baseline week 0, week1, week 2, week 3, week 4 and week 6; and 30 minutes before and 60 minutes after acupuncture through study completion).

ELIGIBILITY:
Inclusion Criteria:

1. aged 20~70 years,
2. met the diagnostic criteria of insomnia according to the Diagnostic and Statistical Manual of Mental Disorders (Fifth Edition, DSM-V)
3. experienced insomnia at least three times a week for more than a month
4. voluntarily agreed with the investigation and signed a written informed con- sent form before the clinical trial started.

Exclusion Criteria:

1. a pregnant or lactating woman
2. the patient's insomnia is caused by mental disorders other than mild anxiety,
3. the patient has serious cardiovascular, liver, kidney or hematopoietic system disease
4. the patient's insomnia is caused by nervous system disease (eg, stroke, Parkinson's Disease)
5. the patient has taken Chinese herbs and herbal formulas for insomnia two weeks before the trial
6. the patient with cardiac pacemaker
7. the patient does not want to wear portable physiological signal recording device (SOMNOwatchTM) and handheld ECG monitor
8. the patient has a history of sleep apnea

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2020-08-07 (Actual); Primary Completion 2021-05-31 (Estimated); Study Completion 2021-08-31 (Estimated)

PRIMARY OUTCOMES:
Changes of The Epworth sleepiness scale (ESS) | Baseline week 0, week 2, week 4 & 2 weeks post-tx (week 6)
  The Epworth sleepiness scale (ESS) containing eight items that ask for self-reported disclosure of the expectation of "dozing" in a variety of situations. A sum of responses is calculated for a total score ranging from 0 to 24, higher scores mean a worse. outcome.
Changes of The HADS(The Hospital Anxiety and Depression Scale) | Baseline week 0, week 2, week 4 & 2 weeks post-tx (week 6)
  The Hospital Anxiety and Depression Scale is a 14-items self-administered questionnaire, the scores ranged from 0 to 21 for anxiety and 0 to 21 for depression, higher scores mean a worse outcome.
Changes of The PSQI(Pittsburgh Sleep Quality Index) | Baseline week 0, week 2, week 4 & 2 weeks post-tx (week 6)
  The 19 questions are combined into seven clinically-derived component scores, each weighted equally from 0-3. The seven component scores are added to obtain a global score ranging from 0-21, with higher scores indicating worse sleep quality.

SECONDARY OUTCOMES:
HRV(Heart rate viability) | Baseline week 0, week1, week 2, week 3, week 4 and week 6; and 30 minutes before and 60 minutes after acupuncture through study completion, an average of 1 year.
  Frequency-domain analysis of heart rate variability (HRV), a noninvasive method, has been used to reflect cardiac autonomic nervous activity in humans. The high-frequency power (HF; 0.15-0.4 Hz) of HRV represents vagal (parasympathetic) control of heart rate. The low-frequency power (LF; 0.04- 0.15 Hz) of HRV is jointly contributed by both sympathetic and vagal nerves, whereas normalized LF (nLF) is regarded as the sympathetic modulation.
actigraphy (3-day) | Baseline week 0, week 2, week 4 & 2 weeks post-tx (week 6)
  Actigraphy provides objective estimates of sleep parameters including: SE(sleep efficiency), SA(sleep awakenings), TST(total sleep time)
sleep diary | Baseline week 0, week 2, week 4 & 2 weeks post-tx (week 6)
  The sleep diary provides daily subjective estimates of sleep parameters including: daytime nap, sleep aids intake, bedtime, sleep onset latency, frequency of nocturnal awakenings, awakenings duration, wake-up time, arising time, feeling upon arising (five-point scale) and sleep quality (five-point scale).

CONTACTS AND LOCATIONS:
Overall Officials: Lee Tsai-Jean, MD, Principal Investigator — Chang Gung Memorial Hospital
Locations (1):
- Chang Gung Memorial Hospital, Keelung, Taiwan

IPD SHARING:
Plan to Share IPD: No
There will be a research number representing the identity. This number will not display the name, identification number, and address.
  For the results and diagnosis of the visit, the research host will maintain a confidential attitude and carefully maintain the privacy. If research results are published, the identity will remain confidential.
  Please also understand that if the participant signs the consent form, the participant agrees that the visit record can be directly reviewed by the monitor, auditor, research ethics committee and the competent authority to ensure that the research process and data comply with relevant laws and regulations.
  These people also promise not to violate the confidentiality of your identity.